CLINICAL TRIAL: NCT06445296
Title: Acute Effects of Animal Versus Plant-Based Protein Within a Realistic High-Fat Meal on Metabolic and Inflammatory Factors
Brief Title: Postprandial Effects of Animal Versus Plant-Based Protein
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ball State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 2103201
Record Dates: First submitted 2024-04-26; First posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-05

CONDITIONS: Overweight or Obesity
Keywords: Plant-based meat alternatives
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant
Masking Description: While complete blinding is not possible (participants will see/taste the food they eat), the investigators will not tell participants whether they are consuming beef or Beyond Meat.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meal Consumption with Beyond Meat (Experimental): During the Beyond Meat arm, participants will consume a high-fat meal containing Beyond Meat (rather than beef). Meals will be otherwise identical.
  Interventions: Other: High-fat meal containing Beyond Meat
- Meal Consumption with Beef (Active Comparator): During the Beef arm, participants will consume a high-fat meal containing beef (rather than Beyond Meat). Meals will be otherwise identical.
  Interventions: Other: High-fat meal containing beef

INTERVENTIONS:
Other: High-fat meal containing beef — High-fat meal (eggs cooked in butter, croissant) with 80% ground beef.
  Arms: Meal Consumption with Beef
Other: High-fat meal containing Beyond Meat — High-fat meal (eggs cooked in butter, croissant) with Beyond Meat Cookout Classic.
  Arms: Meal Consumption with Beyond Meat

SUMMARY:
Shifting away from diets high in animal products towards more plant predominant diets is recommended by many health organizations to both reduce the negative environmental impacts of animal agriculture and to improve health outcomes. As a result, a number of plant-based meat alternatives such as Beyond Meat have been formulated to promote increased plant consumption. However, evidence is limited on the impact of newer plant-based meat alternatives on common cardiometabolic risk factors. The investigators aim to compare the acute metabolic, gastrointestinal, and inflammatory effects of a plant-based meat alternative (i.e., Beyond Meat) versus a comparable beef product within the context of high-fat, "Western-style" meal (i.e., eggs, meat, refined bread product). The investigators will also examine whether these responses differ based on whether individuals have a normal-weight or have overweight/obesity.

DETAILED DESCRIPTION:
The investigators will recruit individuals with a BMI in the normal (18.5-24.9 kg/m2) or overweight/ obesity (>25.0 kg/m2) ranges from the Ball State University campus and surrounding communities. Each participant will complete two meal trials in a randomized crossover design. At each meal trial, a intravenous catheter will be inserted and baseline blood sample collected. Next, participants will consume a high-fat, Western style meal consisting of eggs cooked in butter, a croissant and either 4 oz of 80% ground beef or 4 oz of Beyond Meat ("Cookout Classic" variety). The Beyond Meat and beef products have nearly identical macronutrient profiles, allowing for examination of the unique properties of the two protein sources. Regardless of primary protein source (beef or Beyond Meat), each meal will contain 980 calories (60g fat). Following completion of each meal, blood samples will also be collected 1-, 2-, 3-, and 4-hours. The investigators will measure metabolic markers (i.e., triglycerides, glucose, HDL-C) immediately upon sample collection using the Piccolo Xpress clinical chemistry analyzer. Additional blood will be collected and stored as serum in order to measure indicators of inflammation (e.g., IL-6) and intestinal permeability (e.g., lipopolysaccharide binding protein) using commercially available ELISAs.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 50 years.
* Body mass index > 18.5 kg/m2
* Not pregnant (females only)
* Not postmenopausal (females only).
* Not been diagnosed with cardiovascular disease.
* Not been diagnosed with a cardiometabolic conditions (e.g., type 2 diabetes)
* Not been diagnosed with a chronic inflammatory condition (e.g., rheumatoid arthritis, inflammatory bowel disease).
* Does not regularly take anti-inflammatory drugs (more than 2x week).
* Does not use glucose-lowering drugs (e.g., metformin)
* Does not use lipid-lowering drugs (e.g., statins)
* Does not use tobacco products or any illicit drugs.
* Does not have a pacemaker.
* Can consume pea products (Beyond Meat is made from pea protein).

Exclusion Criteria:

* Not between the ages of 18-50
* Body mass index < 18.5 kg/m2
* Pregnant (females only)
* Postmenopausal status (females only).
* Been diagnosed with cardiovascular disease.
* Been diagnosed with a cardiometabolic conditions (e.g., type 2 diabetes)
* Been diagnosed with a chronic inflammatory condition (e.g., rheumatoid arthritis, inflammatory bowel disease).
* Regularly take anti-inflammatory drugs (more than 2x week).
* Uses glucose-lowering drugs (e.g., metformin)
* Uses lipid-lowering drugs (e.g., statins)
* Uses tobacco products or any illicit drugs.
* Have a pacemaker.
* Allergic to pea products (Beyond Meat is made from pea protein).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Serum interleukin (IL)-6 | Through study completion, up to 1 year.
  The investigators will measure serum IL-6 at baseline and 1-, 2-, 3-, and 4-hours after each meal containing either beef or Beyond Meat. Serum will be banked from each visit and this measurement will take place upon study completion.
Serum lipopolysaccharide binding protein (LBP) | Through study completion, up to 1 year.
  The investigators will measure serum LBP at baseline and 1-, 2-, 3-, and 4-hours after each meal containing either beef or Beyond Meat. Serum will be banked from each visit and this measurement will take place upon study completion.
Serum soluble CD14 (sCD14) | Through study completion, up to 1 year.
  The investigators will measure serum sCD14 at baseline and 1-, 2-, 3-, and 4-hours after each meal containing either beef or Beyond Meat. Serum will be banked from each visit and this measurement will take place upon study completion.
Serum lipopolysaccharide | Through study completion, up to 1 year.
  The investigators will measure serum lipopolysaccharide at baseline and 1-, 2-, 3-, and 4-hours after each meal containing either beef or Beyond Meat. Serum will be banked from each visit and this measurement will take place upon study completion.
Serum tumor necrosis factor (TNF)-alpha | Through study completion, up to 1 year.
  The investigators will measure serum (TNF)-alpha at baseline and 1-, 2-, 3-, and 4-hours after each meal containing either beef or Beyond Meat. Serum will be banked from each visit and this measurement will take place upon study completion.

SECONDARY OUTCOMES:
Triglycerides | Through study completion, up to 1 year.
  The investigators will measure triglycerides at baseline and 1-, 2-, 3-, and 4-hours after each meal containing either beef or Beyond Meat. These measurements will take place immediately and a complete dataset will be compiled upon study completion.
HDL-C | Through study completion, up to 1 year.
  The investigators will measure HDL-C at baseline and 1-, 2-, 3-, and 4-hours after each meal containing either beef or Beyond Meat. These measurements will take place immediately and a complete dataset will be compiled upon study completion.
Glucose | Through study completion, up to 1 year.
  The investigators will measure glucose at baseline and 1-, 2-, 3-, and 4-hours after each meal containing either beef or Beyond Meat. These measurements will take place immediately and a complete dataset will be compiled upon study completion.

OTHER OUTCOMES:
Body composition | Through study completion, up to 1 year.
  The investigators will measure body composition using bioelectrical impedance (InBody).
Systolic and diastolic pressure | Through study completion, up to 1 year.
  The investigators will measure blood pressure using an automated cuff (Omron).

CONTACTS AND LOCATIONS:
Overall Officials: Bryant Keirns, Principal Investigator — Ball State University
Locations (1):
- Health Professions Building, Ball State University, Muncie, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fruit S, Keirns N, Higgins M, Quirk A, Schifferer J, Romanovich O, Yakos A, Osborne K, Trappe S, Keirns BH. Acute effects of a reformulated plant-based meat alternative compared to beef within a high-fat meal on inflammatory and metabolic factors: a randomized crossover trial. Appl Physiol Nutr Metab. 2025 Jan 1;50:1-11. doi: 10.1139/apnm-2024-0498. PMID 40127469